CLINICAL TRIAL: NCT01375114
Title: The Effects of Ginseng on Cancer-Related Fatigue
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Indena S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-0854; NCI-2011-01127 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Results first posted 2023-09-22 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Advanced Cancers; Solid Tumors
Keywords: Advanced Cancers; Solid Tumors; Cancer related fatigue; CRF; Panax ginseng; Placebo; Sugar pill; Functional Assessment of Chronic Illness Therapy-Fatigue; FACIT-F; Quality of life; QOL; FACT-G; Hospital Anxiety and Depression Inventory; Neurocognitive function; SDMT; Global Symptom Evaluation; GSE
MeSH Terms: interventions — Asian ginseng; Sugars; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Panax Ginseng (Experimental): Panax ginseng 400 mg by mouth twice a day from Day 1-29 for first 30 participants in Part 1. Completion of questionnaires taking about 30 minutes on Day 15 (± 3 days), Day 29 (± 3 days), and Day 57 (± 3 days), regarding symptoms such as fatigue, mood, depression, anxiety, nausea, appetite problems, sleep problems, and overall sense of well-being.
  Interventions: Drug: Panax Ginseng; Behavioral: Questionnaires
- Ginseng (Part 2) (Experimental): Panax ginseng 400 mg by mouth twice a day from Day 1-29. Completion of questionnaires taking about 30 minutes on Day 15 (± 3 days), Day 29 (± 3 days), and Day 57 (± 3 days), regarding symptoms such as fatigue, mood, depression, anxiety, nausea, appetite problems, sleep problems, and overall sense of well-being.
  Interventions: Drug: Panax Ginseng; Behavioral: Questionnaires
- Placebo (Part 2) (Placebo Comparator): Oral placebo twice daily for 4 weeks. Completion of questionnaires taking about 30 minutes on Day 15 (± 3 days), Day 29 (± 3 days), and Day 57 (± 3 days), regarding symptoms such as fatigue, mood, depression, anxiety, nausea, appetite problems, sleep problems, and overall sense of well-being.
  Interventions: Dietary Supplement: Placebo; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Panax Ginseng — 400 mg by mouth twice daily from Day 1-29.
  Arms: Ginseng (Part 2); Panax Ginseng
Dietary Supplement: Placebo — Placebo by mouth twice daily for 4 weeks.
  Other Names: Sugar Pill
  Arms: Placebo (Part 2)
Behavioral: Questionnaires — Completion of questionnaires taking about 30 minutes on Day 15 (± 3 days), Day 29 (± 3 days), and Day 57 (± 3 days), regarding symptoms such as fatigue, mood, depression, anxiety, nausea, appetite problems, sleep problems, and overall sense of well-being.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn if panax ginseng (commonly called ginseng) can help to control fatigue and other symptoms such as depression, anxiety, and mood changes in patients with cancer. The safety of ginseng will also be studied.

DETAILED DESCRIPTION:
The Study Supplement:

Ginseng is an herbal supplement that may affect people's energy level, especially during times of fatigue or stress. Many people have used ginseng, but its level of effectiveness and safety has not been clearly studied. In this study, researchers will use questionnaires and other tests to study how ginseng may affect cancer-related fatigue.

Study Groups and Study Drug Administration:

If you are found to be eligible to take part in this study, you will be assigned to a dose of the study drug(s), depending on when you join the study. The first 30 participants will take part in Part 1 of the study. Participants in Part 1 will take ginseng by mouth, in capsule form, every day for 29 days. You will take it 2 times a day (morning and afternoon), and will swallow a total of 2 capsules each day.

If you enroll on this study after the first 30 participants, you will take part in Part 2 of the study. Participants in Part 2 will be randomly assigned (as in the flip of a coin) to 1 of 2 groups:

* Group 1 will take a placebo for 29 days. A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect. If you are assigned to this group, you may be able to take ginseng later, in the second part of the study (described below).
* Group 2 will take ginseng for 29 days, as the Part 1 group did.

You will have an equal chance of being assigned to either group. Neither you nor the study staff will know which group you are in. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Both groups in Part 2 will take ginseng or placebo by mouth, every day for 29 days. You will take it 2 times a day (morning and afternoon), 2 capsules each day.

After your Day 29 ginseng or placebo dose, if you tolerated the doses well, the study doctor may decide you can take ginseng from Days 29-57, following the same dosing schedule you had before.

Study Visits:

On Day 15 (± 3 days), Day 29 (± 3 days), Day 36 (+/- 3 days) and Day 57 (± 3 days), you will fill out questionnaires about the symptoms you may be having, such as fatigue, mood, depression, anxiety, nausea, appetite problems, sleep problems, and your overall sense of well-being. This should take about 30 minutes. You will also be asked about any side effects you may be having. You will also perform a medication review. If you cannot come to the clinic on these days, the research nurse will call and ask you the questions over the phone. The strength and stamina of your arm muscle will be measured only if you come to the clinic. It will not be measured if you are contacted over the phone. Blood (about 1 tablespoon) will be drawn for routine tests on Day 15 (± 3 days), Day 29 (± 3 days) and Day 57 (± 3 days).

The 6-minute walk test will be performed on baseline, Day 15 (± 3 days), Day 29 (± 3 days), and Day 57 (± 3 days).

On Day 8 (± 3 days), Day 21 ( +/- 3 days), Day 36 (± 3 days), and Day 43 (± 3 days), the research nurse will call and ask about the symptoms and side effects you may be having. You will also perform a medication review. This should take about 30 minutes.

If you are unable to return to MD Anderson for your routine blood draw, your local doctor can draw the blood and your results will be sent to MD Anderson.

You blood will be drawn weekly if you are taking coumadin to check to see how fast your blood clots. Liver function tests will also be performed every 2 weeks if you have metastasis to your liver or are on medication such as acetaminophen statins.

Length of Participation:

If you are the among the first thirty patients you will be assigned to receive/take ginseng at the beginning of the study for a total 29 days followed by up to 28 days of ginseng, if the study doctor thinks it is in your best interest. If you are not among the first thirty patients you may receive up to 29 days of ginseng/placebo followed by up to 28 days of ginseng, if the study doctor thinks it is in your best interest. Ginseng/placebo will be stopped early if intolerable side effects occur.

If your main doctor for cancer approves, you may take ginseng after Day 57 (outside of the study) if you tolerated it well.

This is an investigational study. Ginseng is commercially available. Giving ginseng to patients with cancer and fatigue is being done for research purposes only.

Up to 158 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with a histological diagnosis of cancer.
2. Rate fatigue on a numerical scale during the previous 24 hours as >/= 4 on a 0 to 10 scale (0 = no fatigue and 10 = worst possible fatigue).
3. Describe fatigue as being present every day for most of the day for a minimum of 2 weeks.
4. Memorial delirium assessment scale </= 13.
5. Are 18 years or older.
6. Hemoglobin level of >/=8 g/dL within 2 weeks of enrollment. If the patient has not had blood drawn for a hemoglobin level in the previous two weeks, one will be performed to determine eligibility. Patients with a hemoglobin level <9g/dL will be evaluated for treatment of anemia.
7. Able to understand and sign the informed consent.
8. No concurrent use of chronic systemic steroids (defined as currently on more than 1 week of treatment).
9. Controlled pain and depression symptoms, if present ( defined as no change in the Morphine equivalent dose of 30% or change in the dose of antidepressant medication in the past 2 weeks)
10. Patients should have a Zubrod </= 2.
11. All patients who are receiving chemotherapy and/or radiation therapy are eligible for study if they have completed at least one cycle of chemotherapy or targeted therapy, or > 1 week of radiation therapy, and if they have been approved to go on study by their primary oncologist. The PI/designated research staff of this study will obtain and document approval from the primary oncologist and principal investigator of the clinical trial in case the patient is on another clinical trial as referenced in the patient's study documents.
12. Negative pregnancy test for women of childbearing potential, as defined by intact uterus and ovaries, and a history of menses within the last 12 months. Pregnancy test to be performed no greater than 14 days prior to consent in study. In cases of women with elevated b-HCG, these candidates will be eligible to participate so long as the level of b-HCG is not consistent with pregnancy. Women of childbearing potential need to be on or use contraception, or be abstinent during the study period. Their male partners must also use contraception (condom) or maintain abstinence. Birth controls specifications: Women who are able to become pregnant must use birth control during the study and for 30 days after the last ginseng/placebo dose. Acceptable forms of birth control include barrier methods (such as condom or diaphragm) with spermicide.

Exclusion Criteria:

1. Major contraindication to ginseng: allergy/hypersensitivity to Panax species or their constituents (history of arrhythmias, agitation, or motor tics, or severe angina pectoris).
2. Currently taking ginseng, methylphenidate or modafinil or have taken it within the previous 10 days.
3. Inability to complete the baseline assessment forms or to understand the recommendations for participation in the study.
4. Currently with a diagnosis of major depression, manic depressive disorder, obsessive-compulsive disorder, or schizophrenia).
5. Symptomatic tachycardia and uncontrolled hypertension (determined to be clinically significant by the PI).
6. Currently receiving phenobarbital, diphenylhydantoin, primidone, phenylbutazone, MAOIs, clonidine and tricyclic antidepressant drugs
7. Uncontrolled diabetes mellitus as defined by a random blood sugar of >200mg/dl not being monitored by their primary care physician.
8. No concurrent full dose anticoagulant therapy. </= 1 mg/day of coumadin for preventing catheter clots allowed.
9. History of hepatitis A, B and C.
10. Women who are nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-10-14 (Actual); Primary Completion 2016-05-15 (Actual); Study Completion 2025-10-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennurajalingam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yennurajalingam S, Tannir NM, Williams JL, Lu Z, Hess KR, Frisbee-Hume S, House HL, Lim ZD, Lim KH, Lopez G, Reddy A, Azhar A, Wong A, Patel SM, Kuban DA, Kaseb AO, Cohen L, Bruera E. A Double-Blind, Randomized, Placebo-Controlled Trial of Panax Ginseng for Cancer-Related Fatigue in Patients With Advanced Cancer. J Natl Compr Canc Netw. 2017 Sep;15(9):1111-1120. doi: 10.6004/jnccn.2017.0149. PMID 28874596
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the outpatient clinics for palliative care, pain management, internal medicine, and oncology at MD Anderson Cancer Center in Houston, Texas who have been diagnosed with cancer and currently undergoing outpatient chemotherapy at the cancer center, and experiencing Cancer Related Fatigue (CRF) with an average intensity of ≥4/10 on the Edmonton Symptom Assessment Scale (ESAS scale, 0-10) during the 24 hours prior to study enrollment.
Pre-assignment Details: A total of 165 patient were enrolled for this protocol. In Phase-l part of the study, 30 pt received Panax Ginseng and 2 patients withdrew consent. For Phase-II part of study, out of 133 participants, 127 participants were randomized. 6 participants were not randomized for this study for various reasons (participant withdrew n=3, withdrawn at oncologist's request n=1 and due to comorbidities n=2).
Groups:
- Phase-I Panax Ginseng (Single Group); Phase-II Blinded Panax Ginseng: Took one Panax Ginseng capsule (400mg) twice daily by mouth for 29 days
- Phase-ll Blinded Placebo: Took similar appearance colored Placebo capsule twice daily by mouth for 29 days
Period: Overall Study
Arm/Group | Phase-I Panax Ginseng (Single Group) | Phase-II Blinded Panax Ginseng | Phase-ll Blinded Placebo
Started | 30 | 63 | 64
Completed | 24 | 56 | 56
Not Completed | 6 | 7 | 8
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Disease Progression | 3 | 2 | 2
Not completed — Patient Changed Mind | 0 | 0 | 2
Not completed — Pruritus | 0 | 0 | 1
Not completed — Restlessness | 0 | 0 | 1
Not completed — Diarrhea | 0 | 0 | 1
Not completed — Pt enrolled in another clinical trial | 0 | 1 | 0
Not completed — Nausea | 0 | 1 | 0
Not completed — Increased AST/ALT | 0 | 1 | 0
Not completed — Vaginal Hemorrhage | 0 | 1 | 0
Not completed — Family problem | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase-I Panax Ginseng (Single Group) | Phase-II Blinded Panax Ginseng | Phase-ll Blinded Placebo | Total
Number analyzed (Participants) | 30 | 63 | 64 | 157
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [48.0 to 68.0] | 61 [54.0 to 67.0] | 61 [53.3 to 66.8] | 60 [53.0 to 67.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 29 | 24 | 67
  Male | 16 | 34 | 40 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 10 | 1 | 11
  Not Hispanic or Latino | 30 | 53 | 63 | 146
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 6 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 3 | 11
  White | 26 | 59 | 55 | 140
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 63 | 64 | 157

OUTCOME MEASURES:

1. Primary Outcome: Functional Assessment of Chronic Illness Therapy- Fatigue (FACIT-F) Subscale Score Change
Description: "The FACIT-F fatigue subscale was used as the primary outcome measure. There are 13 items in this fatigue subscale. Using the subscale, patients rate the intensity of their fatigue and its related symptoms on a scale of 0 to 4. The total score ranges between 0 and 52, with higher scores denoting less fatigue. The objective was to determine whether the average improvement in FACIT-F fatigue from baseline to Day 29 in patients who received PG was greater than in those who received placebo. We used chi-square test to determine the p-value."
Time Frame: Baseline and Day 29
Population: Those who completed 29 days of trials
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Phase-I Panax Ginseng (SingleGroup); Phase-II Blinded Panax Ginseng: Took one capsule (400mg) twice daily for 29 days
- Phase-ll Blinded Placebo: Took similar appearance colored capsule twice daily for 29 days
Arm/Group | Phase-I Panax Ginseng (SingleGroup) | Phase-II Blinded Panax Ginseng | Phase-ll Blinded Placebo
Number analyzed (Participants) | 24 | 56 | 56
score on a scale | 14.2 (17.5) | 7.5 (12.7) | 6.5 (9.9)
Statistical Analysis 1: Comparison: Phase-I Panax Ginseng (SingleGroup) vs Phase-II Blinded Panax Ginseng; Test type: Other; p = 0.67, Chi-squared

2. Secondary Outcome: Edmonton Symptom Assessment System (ESAS) Fatigue Score Change
Description: The ESAS evaluates 10 commonly experienced symptoms, including pain, fatigue, nausea, depression, anxiety, drowsiness, dyspnea, anorexia, sleep disturbance, and impaired feelings of well-being. The severity of ESAS fatigue was rated on a numerical scale of 0 to 10 (0 = no symptom, 10 = worst possible severity). The objective was to determine whether the average improvement in ESAS fatigue from baseline to Day 29 in patients who received PG was greater than in those who received placebo. We used chi-square test to determine the p-value.
Time Frame: Baseline and Day 29
Population: Those who completed 29 days of trials
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase-I Panax Ginseng (SingleGroup) | Phase-II Blinded Panax Ginseng | Phase-ll Blinded Placebo
Number analyzed (Participants) | 24 | 56 | 56
score on a scale | -2.5 (2.2) | -1.9 (2.6) | -2.1 (2.6)
Statistical Analysis 1: Comparison: Phase-I Panax Ginseng (SingleGroup) vs Phase-II Blinded Panax Ginseng; Test type: Other; p = 0.71, Chi-squared

3. Secondary Outcome: Edmonton Symptom Assessment System (ESAS) Pain Score Change
Description: The ESAS evaluates 10 commonly experienced symptoms, including pain, fatigue, nausea, depression, anxiety, drowsiness, dyspnea, anorexia, sleep disturbance, and impaired feelings of well-being. The severity of ESAS pain was rated on a numerical scale of 0 to 10 (0 = no symptom, 10 = worst possible severity). The objective was to determine whether the average improvement in ESAS pain from baseline to Day 29 in patients who received PG was greater than in those who received placebo. We used chi-square test to determine the p-value.
Time Frame: Baseline and Day 29
Population: Those who completed 29 days of trials
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Phase-II Blinded Panax Ginseng: Took one Panax Ginseng capsule(400mg) twice daily by mouth for 29 days
Arm/Group | Phase-I Panax Ginseng (SingleGroup) | Phase-II Blinded Panax Ginseng | Phase-ll Blinded Placebo
Number analyzed (Participants) | 24 | 56 | 56
score on a scale | -0.9 (1.7) | -0.6 (2.0) | -0.1 (3.0)
Statistical Analysis 1: Comparison: Phase-II Blinded Panax Ginseng vs Phase-ll Blinded Placebo; Test type: Other; p = 0.34, Chi-squared

4. Secondary Outcome: Edmonton Symptom Assessment System (ESAS) Depression Score Change
Description: The ESAS evaluates 10 commonly experienced symptoms, including pain, fatigue, nausea, depression, anxiety, drowsiness, dyspnea, anorexia, sleep disturbance, and impaired feelings of well-being. The severity of ESAS depression was rated on a numerical scale of 0 to 10 (0 = no symptom, 10 = worst possible severity). The objective was to determine whether the average improvement in ESAS depression from baseline to Day 29 in patients who received PG was greater than in those who received placebo. We used chi-square test to determine the p-value.
Time Frame: Baseline and Day 29
Population: Those who completed 29 days of trials
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase-I Panax Ginseng (SingleGroup) | Phase-II Blinded Panax Ginseng | Phase-ll Blinded Placebo
Number analyzed (Participants) | 24 | 56 | 56
score on a scale | 0.0 (1.7) | -0.3 (2.2) | 0.1 (2.2)
Statistical Analysis 1: Comparison: Phase-II Blinded Panax Ginseng vs Phase-ll Blinded Placebo; Test type: Other; p = 0.36, Chi-squared

5. Secondary Outcome: Edmonton Symptom Assessment System (ESAS) Drowsiness Score Change
Description: The ESAS evaluates 10 commonly experienced symptoms, including pain, fatigue, nausea, depression, anxiety, drowsiness, dyspnea, anorexia, sleep disturbance, and impaired feelings of well-being. The severity of ESAS drowsiness was rated on a numerical scale of 0 to 10 (0 = no symptom, 10 = worst possible severity). The objective was to determine whether the average improvement in ESAS drowsiness from baseline to Day 29 in patients who received PG was greater than in those who received placebo. We used chi-square test to determine the p-value.
Time Frame: Baseline and Day 29
Population: Those who completed 29 days of trials
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase-I Panax Ginseng (SingleGroup) | Phase-II Blinded Panax Ginseng | Phase-ll Blinded Placebo
Number analyzed (Participants) | 24 | 56 | 56
score on a scale | -0.8 (2.2) | -0.9 (3.1) | -0.6 (3.2)
Statistical Analysis 1: Comparison: Phase-II Blinded Panax Ginseng vs Phase-ll Blinded Placebo; Test type: Other; p = 0.56, Chi-squared

ADVERSE EVENTS:
Time Frame: Baseline up to 57 days
Description: Adverse events that were reported by the patient
Groups:
- Open Label Extension: One capsule 400mg by mouth twice a day for 29 days
Arm/Group | Phase-I Panax Ginseng (Single Group) | Phase-II Blinded Panax Ginseng | Phase-ll Blinded Placebo | Open Label Extension
All-Cause Mortality (participants affected / at risk) | 1/30 | 1/63 | 0/64 | 0/102
Serious Adverse Events (participants affected / at risk) | 3/30 | 2/63 | 1/64 | 0/102
Other Adverse Events (participants affected / at risk) | 4/30 | 6/63 | 5/64 | 9/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase-I Panax Ginseng (Single Group) (N=30) | Phase-II Blinded Panax Ginseng (N=63) | Phase-ll Blinded Placebo (N=64) | Open Label Extension (N=102)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal disorder (Other) (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Breast Infection (Infections and infestations) | 0 | 1 | 0 | 0
White Blood Cell disorder (Investigations) | 1 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase-I Panax Ginseng (Single Group) (N=30) | Phase-II Blinded Panax Ginseng (N=63) | Phase-ll Blinded Placebo (N=64) | Open Label Extension (N=102)
Hyperglycemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Appendicitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Fatigue (Nervous system disorders) | 0 | 0 | 1 | 1
Hypokalemia (Cardiac disorders) | 0 | 0 | 0 | 1
Allergic reaction (Cardiac disorders) | 0 | 0 | 0 | 1
Infections and Infestations (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Thrombotic Thrombocytopenic purpura (Vascular disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral Mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Breast Infection (Infections and infestations) | 0 | 1 | 0 | 0
General disorders (other) (General disorders) | 0 | 1 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Increased ALT (Investigations) | 0 | 1 | 0 | 0
Increased AST (Investigations) | 0 | 1 | 0 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Delirium (Nervous system disorders) | 1 | 0 | 0 | 0
Insomnia (Nervous system disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Chest pain (Cardiac disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT01375114/Prot_SAP_000.pdf